Improving Health and Employment Outcomes Through Workplace Opioid Policies NCT05387408

Human Subjects Approval: 08/05/2022

FOR IRB USE ONLY IRB ID #: 202205011 APPROVAL DATE: 05/05/22 RELEASED DATE: 05/05/22 EXPIRATION DATE: N/A

We invite you to participate in a research study being conducted by Dr. Ann Marie Dale from Washington University in St. Louis. The purpose of this study is to evaluate a union and health fund's use of guidelines to reduce opioid misuse among their members. We are seeking workers to complete this survey to evaluate the use of the guidelines.

If you choose to participate, you will be a volunteer for the study; you will be asked to complete a 10 minute survey; and you may skip any questions that you prefer not to answer. All information will be anonymous. We will not ask any questions that identify you. The survey questions ask about your knowledge of health benefits and policies, attitudes toward use of opioid prescriptions, and participation in union programs and benefits.

There are no known risks and no costs to you for participation. You will not be penalized or lose any benefits for which you otherwise qualify and participation will not affect your job. There is no compensation for participation. Although you will not directly benefit from participation, your information may help improve health risks of others in the construction industry. If you choose not to participate, please do not answer any of the questions and exit out of this webpage. Your data will be stored without your name or any other information that would allow us to identify you. Your data may be used in future research studies and cannot be removed. By allowing us to use your data you give up any property rights you may have in the data. We will share your data with a large data repository (a repository is a database of information) for use by the research community. Your individual identify will not be known in this data set.

If you have any questions about the research study itself, please contact: Sam Biver at sbiver@wustl.edu. If you feel you have been harmed from being in the study, please contact: Dr. Ann Marie Dale at amdale@wustl.edu. If you have questions, concerns, or complaints about your rights as a research participant, please contact the Human Research Protection Office at 1-(800)-438-0445 or email hrpo@wustl.edu. General information about being a research participant can be found on the Human Research Protection Office web site, http://hrpo.wustl.edu. Thank you very much for your consideration of this research study.